CLINICAL TRIAL: NCT06909344
Title: Effectiveness and Safety of 577-nm Diode Laser in the Treatment of Non -Inflammatory Acne
Brief Title: 577-nm Diode Laser in the Treatment of Non -Inflammatory Acne
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hala Hassan Shehata Ahmed, resident physician at dermatology department at azhar assuit university hospital, Al-Azhar University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yellow laser in comedonal acne
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-02

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- All patients will be treated with sessions of the 577 nm Diode laser on one side of the face (Active Comparator): All patients will be treated with sessions of the 577 nm Diode laser on one side of the face and on the other side serve as a control
  Interventions: Device: 577 nm Diode laser
- other side of the face serve as a control arm without interventions (No Intervention): All patients will be treated with sessions of the 577 nm Diode laser on one side of the face and on the other side serve as a control without any interventions

INTERVENTIONS:
Device: 577 nm Diode laser — All patients will be treated with sessions of the 577 nm Diode laser on one side of the face and on the other side serve as a control
  Arms: All patients will be treated with sessions of the 577 nm Diode laser on one side of the face

SUMMARY:
The aim of this study is to evaluate the clinical efficacy and safety of the 577 nm diode laser in the treatment of non -inflammatory acne.

DETAILED DESCRIPTION:
Acne vulgaris is a prevalent skin condition categorized into two types: non-inflammatory (comedones) and inflammatory (papules, pustules, and nodules). It primarily affects adolescents and young adults, often leading to scarring and diminished self-esteem. Over 80% of teenagers experience acne, which can continue into adulthood. The psychological impacts are significant, as many individuals experience reduced self-esteem and heightened anxiety. Effective treatment and management are essential for enhancing the quality of life for those affected.

The pathogenesis of acne is influenced by multiple factors, including excess sebum production, follicular keratinization, Propionibacterium acnes colonization, and inflammation. Acne treatments typically include topical and oral medications. Topical options, such as retinoids and antibiotics, require frequent application, which can affect patient compliance. Topical antibiotics often show poor efficacy and can lead to recurrence. Additionally, topical retinoids may cause irritation, while oral medications can have more severe side effects. Systemic isotretinoin is effective but associated with high costs and significant side effects, including teratogenicity and dryness.

Laser treatment for acne, particularly the inflammatory type, has gained significant popularity in recent years. This therapy effectively reduces acne lesions by inhibiting overactive sebaceous glands and alleviating inflammation. The mechanism is believed to involve the activation of porphyrins produced by Propionibacterium acnes, leading to the destruction of their cell membranes. Lasers with a wavelength of 1064 nm have been specifically studied for acne treatment. Various laser systems, such as near-infrared lasers and radiofrequency devices, effectively destroy sebaceous glands. Additionally, light sources like blue lights and intense pulsed light (IPL) are being increasingly incorporated into standard medical treatments to improve therapeutic outcomes.

Several types of lasers have been used to treat acne vulgaris in recent years and have shown great results. IPL and the 1,064-nm Nd:YAG laser are effective in treating inflammatory facial acne vulgaris, with no significant difference in their effects on facial acne lesions. Nd:YAG laser treatment also leads to a reduction in the total number of comedones, similar to the improvement observed with inflammatory lesions.

Vascular lasers, particularly a 577-nm high-power optically pumped semiconductor laser, are effective and safe for treating inflammatory lesions, decreasing Propionibacterium acnes, and reducing the size and function of the pilosebaceous unit.

Effective management of acne comedones often requires consistent use of topical treatments for several weeks to see significant improvement. If over-the-counter options take a long time and require considerable effort, it may be beneficial to explore other therapeutic avenues.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acne comedones
* Patients' ages range from 18-40 years.
* Minimum 10 comedonal lesions on both half of the face

Exclusion Criteria:

* Patients with systemic disease interfere with healing.
* Patients with Photosensitivity.
* Pregnant or lactating females.
* Previous topical, systemic, laser, surgical treatment and comedogenic drugs in the last 3 months.
* Skin cancer or suspicious lesions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-29 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of comedones, measured through clinical assessment before and after treatment | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Azhar Assuit university hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbieri JS, Spaccarelli N, Margolis DJ, James WD. Approaches to limit systemic antibiotic use in acne: Systemic alternatives, emerging topical therapies, dietary modification, and laser and light-based treatments. J Am Acad Dermatol. 2019 Feb;80(2):538-549. doi: 10.1016/j.jaad.2018.09.055. Epub 2018 Oct 5. PMID 30296534
- [Background] Mavranezouli I, Daly CH, Welton NJ, Deshpande S, Berg L, Bromham N, Arnold S, Phillippo DM, Wilcock J, Xu J, Ravenscroft JC, Wood D, Rafiq M, Fou L, Dworzynski K, Healy E. A systematic review and network meta-analysis of topical pharmacological, oral pharmacological, physical and combined treatments for acne vulgaris. Br J Dermatol. 2022 Nov;187(5):639-649. doi: 10.1111/bjd.21739. Epub 2022 Aug 22. PMID 35789996
- [Background] Melnik BC. Acne Transcriptomics: Fundamentals of Acne Pathogenesis and Isotretinoin Treatment. Cells. 2023 Nov 10;12(22):2600. doi: 10.3390/cells12222600. PMID 37998335
- [Background] Alsohaimi AO, Alghamdi A, Alghamdi RS, Alghamdi AH, Alkhathami AM, Alghamdi MA, Alghamdi SA, Alzahrani NM, Alghamdi NS. Prevalence of Acne Vulgaris in Adolescents and Young Adults in Al-Baha Region, Saudi Arabia. Cureus. 2024 Oct 12;16(10):e71293. doi: 10.7759/cureus.71293. eCollection 2024 Oct. PMID 39529772
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK459173/